CLINICAL TRIAL: NCT00381680
Title: Intensive Treatment for Intermediate-Risk Relapse of Childhood B-precursor Acute Lymphoblastic Leukemia (ALL): A Randomized Trial of Vincristine Strategies
Brief Title: Low-Dose or High-Dose Vincristine and Combination Chemotherapy in Treating Young Patients With Relapsed B-Cell Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AALL0433; NCI-2009-00306 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-AALL0433 (Other: Children's Oncology Group); CDR0000495359 (Other: Clinical Trials.gov); U10CA098543 (NIH)
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: B-cell Childhood Acute Lymphoblastic Leukemia; L1 Childhood Acute Lymphoblastic Leukemia; L2 Childhood Acute Lymphoblastic Leukemia; Intermediate Risk Recurrent Childhood Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Vincristine; Prednisone; Doxorubicin; pegaspargase; Cytarabine; Methotrexate; merphos; Dexamethasone; Calcium Dobesilate; Etoposide; Cyclophosphamide; Leucovorin; Filgrastim; Granulocyte Colony-Stimulating Factor; Asparaginase; palmitoyl-L-asparaginase; Mercaptopurine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regimen A: Standard vincristine dosing (Active Comparator): See detailed description.
  Interventions: Drug: vincristine sulfate; Drug: prednisone; Drug: doxorubicin hydrochloride; Drug: pegaspargase; Drug: cytarabine; Drug: methotrexate; Drug: dexamethasone; Drug: etoposide; Drug: cyclophosphamide; Drug: leucovorin calcium; Biological: filgrastim; Drug: asparaginase; Drug: mercaptopurine
- Arm B: Randomized High Dose Vincristine regimen (Experimental): See detailed description. Closed to accrual as of 09/2010).
  Interventions: Drug: vincristine sulfate; Drug: prednisone; Drug: doxorubicin hydrochloride; Drug: pegaspargase; Drug: cytarabine; Drug: methotrexate; Drug: dexamethasone; Drug: etoposide; Drug: cyclophosphamide; Drug: leucovorin calcium; Biological: filgrastim; Drug: asparaginase; Drug: mercaptopurine

INTERVENTIONS:
Drug: vincristine sulfate — Given IV
  Other Names: leurocristine sulfate; VCR; Vincasar PFS
Drug: prednisone — Given PO
  Other Names: DeCortin; Deltra
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: pegaspargase — Given IM
  Other Names: L-asparaginase with polyethylene glycol; Oncaspar; PEG-ASP; PEG-L-asparaginase
Drug: cytarabine — Given IT or IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Drug: methotrexate — Given IT or IV
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
Drug: dexamethasone — Given PO
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: leucovorin calcium — Given IV or PO
  Other Names: CF; CFR; LV
Biological: filgrastim — Given IV or SC
  Other Names: G-CSF; Neupogen
Drug: asparaginase — Given IM
  Other Names: ASNase; Colaspase; Crasnitin; Elspar; L-ASP
Drug: mercaptopurine — Given PO
  Other Names: 6-mercaptopurine; 6-MP; Leukerin; MP

SUMMARY:
This randomized phase III trial is studying low-dose vincristine to see how well it works compared with high-dose vincristine when given together with different combination chemotherapy regimens in treating young patients with intermediate-risk relapsed B-cell acute lymphoblastic leukemia. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) and giving the drugs in different ways and different doses may kill more cancer cells..

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the efficacy of an intensive chemotherapy regimen (based on POG-9412) for pediatric patients with intermediate-risk relapsed B-precursor acute lymphoblastic leukemia.

SECONDARY OBJECTIVES:

I. To determine levels of minimal residual disease (MRD) present at the end of the first & third blocks of Induction and determine if higher MRD levels at these times identify patients at higher risk of relapse who might be candidates for alternative therapies in future trials.

II. To determine whether common polymorphisms in candidate genes are associated with the frequency of vincristine adverse effects (peripheral neuropathy, syndrome of inappropriate antidiuretic hormone secretion [SIADH], or constipation) and with anti-leukemic response (level of end-Induction MRD).

III. Compare, descriptively, the outcomes of patients treated with combination chemotherapy vs those treated with matched sibling-related donor hematopoietic stem cell transplantation (for those with eligible donors).

IV. To use deoxyribonucleic acid (DNA) arrays to characterize patterns of gene expression that predict treatment failure, and to compare gene expression profiles at the time of relapse with those at initial diagnosis to gain an understanding of the pathways that may be involved in disease resistance.

OUTLINE: This is a multicenter, randomized study. Patients are randomized to 1 of 2 treatment regimens (randomization closed as of 09/2010).

INDUCTION THERAPY 1 (WEEKS 1-5):

Regimen A: Patients receive low-dose vincristine intravenously (IV) on days 1, 8, 15, and 22; prednisone orally (PO) 3 times daily (TID) on days 1-28; doxorubicin hydrochloride IV over 15 minutes on day 1; pegaspargase intramuscularly (IM) on days 2, 8, 15, and 22; cytarabine intrathecally (IT) on day 1; and methotrexate IT* on days 15 and 29.

Regimen B: (closed to accrual as of 09/2010)***: Patients receive high-dose vincristine IV on days 1, 8, 15, and 22 and prednisone, doxorubicin hydrochloride, pegaspargase, cytarabine, and methotrexate* as in Regimen A.

NOTE: *Central nervous system (CNS)-positive patients do not receive methotrexate IT. In both arms, CNS-positive patients receive intrathecal triple therapy (ITT) comprising methotrexate IT, hydrocortisone IT, and cytarabine IT on days 1, 8, 15, 22, and 29. CNS-positive patients not achieving remission after induction therapy 1 receive one additional dose of ITT on day 36. Patients in both arms then proceed to induction therapy 2**.

NOTE: **Patients who are CNS-positive at relapse receive induction therapy 3 BEFORE induction therapy 2.

NOTE: ***Patients already enrolled on Regimen B are crossover to Regimen A.

INDUCTION THERAPY 2 (WEEKS 6-10 or 7-11): Once blood counts recover, all patients receive etoposide phosphate IV over = 1 hour and cyclophosphamide IV over 1 hour on days 1-5; high-dose methotrexate IV continuously over 24 hours on day 22; leucovorin calcium IV or PO beginning 42 hours after start of high-dose methotrexate and continuing every 6 hours for at least 3 doses; and methotrexate IT* on days 1 and 22. Patients also receive filgrastim (G-CSF) IV or subcutaneously (SC) beginning on day 6 and continuing until blood counts recover.

NOTE: *CNS-positive patients do not receive methotrexate IT. CNS-positive patients receive ITT on days 1 and 22. Patients with testicular-relapse with persistent testicular disease at the end of induction therapy 1 undergo testicular radiotherapy once daily (QD), 5 days a week, for 12 days during induction therapy 2**.

NOTE: **Radiotherapy should be completed before beginning high-dose methotrexate (week 9) chemotherapy.

All patients then proceed to induction therapy 3.

INDUCTION THERAPY 3 (WEEKS 11-15 or 12-16): All patients receive high-dose cytarabine IV over 3 hours on days 1, 2, 8, and 9, and asparaginase IM on days 2 and 9. Patients also receive G-CSF IV or SC beginning on day 10 and continuing until blood counts recover. Patients with a suitable HLA-matched related donor are removed from study and proceed to stem cell transplantation. Patients without a suitable HLA-matched related donor proceed to intensification therapy 1 (as per their randomized regimen in induction therapy 1).

INTENSIFICATION THERAPY 1 (WEEKS 16-27 or 17-28):

Regimen A: Patients receive low-dose vincristine IV and high-dose methotrexate IV continuously over 24 hours on day 1; leucovorin calcium IV or orally beginning 42 hours after start of high-dose methotrexate and continuing every 6 hours for at least 3 doses; oral mercaptopurine once daily on days 2-6; etoposide phosphate IV over ≥ 1 hour and cyclophosphamide IV over 1 hour on day 8; and methotrexate IT* on day 15. Treatment repeats every 21 days for 4 courses (with the exception of IT methotrexate which repeats for only 3 courses).

Regimen B: Patients receive high-dose vincristine IV on day 1 and high-dose methotrexate, leucovorin calcium, mercaptopurine, etoposide phosphate, cyclophosphamide, and methotrexate IT* as in Regimen A. (closed to accrual as of 09/2010)

NOTE: *CNS-positive patients do not receive methotrexate IT. CNS-positive patients receive ITT on day 15. ITT repeats every 3 weeks for 3 courses.

NOTE: ** Patients already enrolled on Regimen B are crossover to Regimen A.

Patients in both regimens then proceed to reinduction therapy (as per their randomized regimen in induction therapy 1).

REINDUCTION THERAPY (WEEKS 28-32 or 29-33):

Regimen A: Patients receive low-dose vincristine IV and doxorubicin hydrochloride IV over 15 minutes on days 1, 8, and 15, oral dexamethasone twice daily on days 1-7 and 15-21, pegaspargase IM on days 2 and 15, and methotrexate IT* on days 1 and 28.

Regimen B: Patients receive high-dose vincristine IV on days 1, 8, and 15 and doxorubicin hydrochloride, dexamethasone, pegaspargase, and methotrexate IT* as in Regimen A. (closed to accrual as of 09/2010)

NOTE: *CNS-positive patients do not receive methotrexate IT. CNS-positive patients receive ITT on days 1 and 28.

NOTE: ** Patients already enrolled on Regimen B are crossover to Regimen A. Patients in both regimens then proceed to intensification therapy 2 (as per their randomized regimen in induction therapy 1).

INTENSIFICATION THERAPY 2 (WEEKS 33-56 or 34-57):

Regimen A: Once blood counts recover, patients receive high-dose cytarabine IV over 3 hours on days 1 and 2; pegaspargase IM on day 2; low-dose vincristine IV on days 22 and 29; high-dose methotrexate IV on day 22; leucovorin calcium IV or orally beginning 42 hours after start of high-dose methotrexate and continuing every 6 hours for at least 3 doses; oral mercaptopurine once daily on days 23-27; etoposide phosphate IV over ≥ 1 hour and cyclophosphamide IV over 1 hour on day 29; and methotrexate IT* on day 36. Patients also receive G-CSF IV or SC beginning on day 3 and continuing until blood counts recover. Treatment repeats every 42 days for 4 courses (with the exception of IT methotrexate which only repeats for 3 courses).

Regimen B: Patients receive high-dose cytarabine, high-dose methotrexate, leucovorin calcium, pegaspargase, mercaptopurine, etoposide phosphate, cyclophosphamide, methotrexate IT*, and G-CSF as in Regimen A. Patients also receive high-dose vincristine IV on days 22 and 29.

NOTE: *CNS-positive patients do not receive methotrexate IT. CNS-positive patients receive ITT on day 36. Treatment repeats every 6 weeks for 3 courses.

Patients in both regimens then proceed to maintenance therapy (as per their randomized regimen in induction therapy 1).

MAINTENANCE THERAPY (week 57-106 or 58-107):

Regimen A: Patients receive methotrexate IT on day 1* and then PO on days 8, 15, 22, 29, and 36; mercaptopurine PO QD on days 1-42; dexamethasone PO twice daily (BID) on days 1-5; and low-dose vincristine IV and cyclophosphamide IV over 1 hour on days 43, 50, 57, and 64. Treatment repeats every 70 days for 5 courses.

Regimen B: Patients receive methotrexate*, mercaptopurine, dexamethasone, and cyclophosphamide as in Regimen A. Patients also receive high-dose vincristine IV on days 43, 50, 57, and 64.

NOTE: *CNS-positive patients receive methotrexate IT on day 1, instead of oral methotrexate.

Beginning in week 1 of the first maintenance therapy course, patients with CNS relapse undergo cranial radiotherapy QD, 5 days a week, for 10 days. Patients with CNS relapse do not receive any IT therapy during maintenance therapy.

After completion of study therapy, patients are followed periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute lymphoblastic leukemia (ALL)

  * Bone marrow with > 25% L1 or L2 lymphoblasts (M3 marrow)

    * Patients with > 25% L3 marrow lymphoblasts and/or evidence of c-myc translocation are not eligible (considered Burkitt's or mature B-cell leukemia)
* Intermediate-risk relapsed disease, meeting 1 of the following criteria:

  * Bone marrow relapse ≥ 36 months after initial diagnosis (defined as M3 marrow after previous remission from ALL)
  * Combined bone marrow and extramedullary (CNS* and/or testicular**) relapse ≥ 36 months after initial diagnosis
  * Isolated extramedullary (CNS* and/or testicular**) relapse < 18 months after initial diagnosis
* The following subtypes are not allowed:

  * T-lineage ALL
  * Mature B-cell (Burkitt's) leukemia (defined as L3 morphology and/or evidence of c-myc translocation)
  * Philadelphia-chromosome positive disease
* No Down syndrome (trisomy 21)
* Shortening fraction >= 27% by echocardiogram OR ejection fraction >= 50% by radionuclide angiogram
* Bilirubin < 3.0 mg/dL
* Not pregnant
* Fertile patients must use effective contraception
* No history of peripheral neuropathy >= grade 3 within the past month
* No toxicity (i.e. peripheral neuropathy) >= grade 3 attributable to vincristine within the past month
* At least 5 days since prior intrathecal chemotherapy
* No prior hematopoietic stem cell or marrow transplantation
* No prior cranial radiotherapy > 1200 cGy (for patients with CNS relapse)
* No concurrent stem cell transplant
* No concurrent alternative therapy
* No concurrent itraconazole in patients receiving vincristine
* No concurrent intensity-modulated radiotherapy

Ages: 1 Year to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 275 (Actual)
Dates: Start 2007-03; Primary Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glen Lew, MD, Principal Investigator — Children's Oncology Group
Locations (173):
- United States (159):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Children's Oncology Group, Arcadia, California
  - Southern California Permanente Medical Group, Downey, California
  - City of Hope Medical Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's Hospital, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Childrens Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter General Hospital, Sacramento, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - University of California San Francisco Medical Center-Parnassus, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lombardi Comprehensive Cancer Center at Georgetown University, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - University of Florida, Gainesville, Florida
  - Nemours Children's Clinic - Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Florida Hospital, Orlando, Florida
  - M D Anderson Cancer Center- Orlando, Orlando, Florida
  - Nemours Childrens Clinic - Orlando, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph Children's Hospital of Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Georgia Regents University, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii, Honolulu, Hawaii
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - University of Illinois, Chicago, Illinois
  - Childrens Memorial Hospital, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Hope Children's Hospital, Oak Lawn, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Services, Indianapolis, Indiana
  - Raymond Blank Children's Hospital, Des Moines, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Children's Hospital-Main Campus, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Michigan State University - Breslin Cancer Center, Lansing, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri-Columbia, Columbia, Missouri
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - UMDNJ - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - New York University Langone Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospitals Inc, Asheville, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Hospital, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Children's Medical Center of Dayton, Dayton, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Palmetto Health Richland, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Science Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Childrens Hospital-King's Daughters, Norfolk, Virginia
  - Carilion Clinic Children's Hospital, Roanoke, Virginia
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston, Charleston, West Virginia
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (11):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Chedoke-McMaster Hospitals, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital Sainte-Justine, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Switzerland (2):
  - Swiss Pediatric Oncology Group - Bern, Bern
  - Swiss Pediatric Oncology Group - Lausanne, Lausanne

IPD SHARING:
Plan to Share IPD: Yes
Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive

REFERENCES:
- [Derived] Lew G, Chen Y, Lu X, Rheingold SR, Whitlock JA, Devidas M, Hastings CA, Winick NJ, Carroll WL, Wood BL, Borowitz MJ, Pulsipher MA, Hunger SP. Outcomes after late bone marrow and very early central nervous system relapse of childhood B-acute lymphoblastic leukemia: a report from the Children's Oncology Group phase III study AALL0433. Haematologica. 2021 Jan 1;106(1):46-55. doi: 10.3324/haematol.2019.237230. PMID 32001530
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Regimen A: Standard Vincristine Dosing: Standard VCR dosing (1.5 mg/m^2, max 2 mg)
- Regimen B: Randomized High Dose Vincristine Regimen: Intensive VCR dosing (2 mg/m^2, max 2.5 mg)
Period: Overall Study
Arm/Group | Regimen A: Standard Vincristine Dosing | Regimen B: Randomized High Dose Vincristine Regimen
Started | 206 | 69
Completed | 81 | 19
Not Completed | 125 | 50
Not completed — Adverse Event | 9 | 3
Not completed — Death | 10 | 7
Not completed — Lost to Follow-up | 3 | 2
Not completed — Physician Decision | 25 | 6
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Entry onto another COG Trial | 1 | 2
Not completed — Alternative Therapy | 11 | 5
Not completed — Secondary Malignancy | 3 | 0
Not completed — Delay initiation | 1 | 0
Not completed — Stem Cell Transplant | 26 | 10
Not completed — Relapse | 18 | 9
Not completed — Induction Failure | 4 | 1
Not completed — Progression | 1 | 1
Not completed — Other not otherwise specified | 7 | 2
Not completed — Ineligible | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm B: Randomized High Dose Vincristine Regimen: Intensive VCR dosing (2 mg/m^2, max 2.5 mg)
- Total: Total of all reporting groups
Arm/Group | Regimen A: Standard Vincristine Dosing | Arm B: Randomized High Dose Vincristine Regimen | Total
Number analyzed (Participants) | 206 | 69 | 275
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.21 (5.20) | 19.62 (4.84) | 17.82 (5.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 25 | 121
  Male | 110 | 44 | 154
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 55 | 8 | 63
  Not Hispanic or Latino | 145 | 51 | 196
  Unknown or Not Reported | 6 | 10 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 12 | 3 | 15
  White | 157 | 55 | 212
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 28 | 9 | 37

OUTCOME MEASURES:

1. Primary Outcome: Event Free Survival. EFS
Description: Percentage of patients who were event free at 3 years among those on Standard VCR dosing who did not undergo Hematopoietic Stem Cell Transplant (SCT).
Time Frame: 3 years after enrollment
Population: The analysis is limited to eligible patients on regimen A (Standard VCR dosing) who did not undergo SCT.
Measure: Number (95% Confidence Interval); unit: percentage of participants EFS at 3 yrs3
Arm/Group | Regimen A: Standard Vincristine Dosing
Number analyzed (Participants) | 142
percentage of participants EFS at 3 yrs3 | 66.0 [58.0 to 74.0]

2. Secondary Outcome: Frequency and Severity of Adverse Effects
Description: Percentage of patients who developed at least 1 episode of grade 2 to 4 neuropathy.
Time Frame: Up to 107 weeks
Population: The total number of patients for CC or CT genotype is 81 and for high-risk CEP72 genotype is 18. No related by arm data were provided.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- All Patients: This analysis looks at all eligible patients with CC or CT genotypes as well as all eligible patients with the high-risk CEP72 genotype (TT at rs924607).
Arm/Group | All Patients
Number analyzed (Participants) | 99
percentage of participants
  CC or CT genotype: number analyzed (Participants) | 81
  CC or CT genotype | 17.3 [10.1 to 27.6]
  High-risk CEP72 genotype (TT at rs924607): number analyzed (Participants) | 18
  High-risk CEP72 genotype (TT at rs924607) | 44.4 [22.4 to 68.7]

3. Secondary Outcome: Gene Expression Profile
Description: Percent of unfavorable gene expression profile of early versus late marrow relapse.
Time Frame: Up to 36 months
Population: The data were not collected due to the lack of funds.
Arm/Group | Regimen A: Standard Vincristine Dosing | Arm B: Randomized High Dose Vincristine Regimen
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Rate of Minimal Residual Disease (MRD) < 0.01% at End Block 1
Description: Percentage of patients who had minimal residual disease (MRD) < 0.01% among those with isolated BM or combined BM relapse >= 36 months and had successful MRD determinations at End Block 1
Time Frame: End of Block 1 (35 days) of Induction therapy
Population: This analysis is limited to all eligible patients with isolated BM or combined BM relapse >= 36 months and had successful MRD determinations at End Block 1.
Measure: Number; unit: percentage of participants
Groups:
- Regimen A: Standard VCR dosing (1.5 mg/m^2, max 2 mg)
- Regimen B: Intensive VCR dosing (2 mg/m^2, max 2.5 mg)
Arm/Group | Regimen A | Regimen B
Number analyzed (Participants) | 122 | 53
percentage of participants | 50.8 | 41.5

5. Secondary Outcome: Rate of Minimal Residual Disease (MRD) < 0.01% at End Block 3
Description: Percentage of patients who had minimal residual disease (MRD) < 0.01% among those with isolated BM or combined BM relapse >= 36 months and had successful MRD determinations at End Block 3.
Time Frame: End of Block 3 (105 days) of Induction therapy
Population: This analysis is limited to all eligible patients with isolated BM or combined BM relapse >= 36 months and had successful MRD determinations at End Block 3.
Measure: Number; unit: percentage of participants
Groups:
- Regimen A: Standard VCR dosing (1.5 mg/m^2, max 2mg)
Arm/Group | Regimen A | Regimen B
Number analyzed (Participants) | 70 | 27
percentage of participants | 81.4 | 88.9

6. Secondary Outcome: Event Free Survival (EFS)
Description: Percentage of patients who were event free at 3 years among those with isolated BM or combined BM relapse >= 36 months.
Time Frame: 3 years
Population: The percentage of patients (pts) who were event free at 3 years among those with isolated BM or combined BM relapse >= 36 months. Pts with MRD <0.01% at the end of Block 1 (MRD < 0.01% BL1); MRD >= 0.01% at the end of Block 1 (MRD>= 0.01% BL1); MRD < 0.01% at the end of Block 3 (MRD < 0.01% BL3);MRD >=0.01% at the end of Block 3.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Regimen A | Regimen B
Number analyzed (Participants) | 127 | 54
percentage of participants
  MRD < 0.01% BL1: number analyzed (Participants) | 62 | 22
  MRD < 0.01% BL1 | 88.5 [80.4 to 96.6] | 77.3 [59.8 to 94.8]
  MRD >= 0.01% BL1: number analyzed (Participants) | 60 | 31
  MRD >= 0.01% BL1 | 60.0 [47.6 to 72.4] | 46.2 [27.8 to 64.7]
  MRD < 0.01% BL3: number analyzed (Participants) | 57 | 24
  MRD < 0.01% BL3 | 83.8 [74.0 to 93.5] | 83.3 [68.4 to 98.2]
  MRD >= 0.01% BL3: number analyzed (Participants) | 13 | 3
  MRD >= 0.01% BL3 | 61.5 [35.1 to 88.0] | 33.3 [0.0 to 86.7]

7. Secondary Outcome: Adjusted Event Free Survival
Description: Adjusted percentage of patients who were event free at 3 years. For patients who received matched donor SCT, EFS was adjusted to start from the actual SCT date. For patients who did not undergo SCT, EFS was adjusted to start from median time to SCT based on patients who received matched related SCT (where patients who had events prior to SCT date were excluded from the calculation of median time to SCT).
Time Frame: 3 years
Population: The analysis is limited to eligible patients on Standard VCR dosing who received matched related SCT, excluding patients who had events prior to receiving SCT. And those patients on Regimen A who did not undergo SCT, excluding patients who went off therapy prior to the adjusted starting time.
Measure: Number (95% Confidence Interval); unit: adjusted percentage of participants
Arm/Group | Regimen A: Standard Vincristine Dosing
Number analyzed (Participants) | 152
adjusted percentage of participants
  Received SCT: number analyzed (Participants) | 34
  Received SCT | 82.2 [68.8 to 95.5]
  Did not receive SCT: number analyzed (Participants) | 118
  Did not receive SCT | 64.2 [55.3 to 73.1]

ADVERSE EVENTS:
Description: Only eligible patients are included in the toxicity adverse events for both serious and other.
Arm/Group | Regimen A: Standard Vincristine Dosing | Arm B: Randomized High Dose Vincristine Regimen
Serious Adverse Events (participants affected / at risk) | 40/203 | 11/68
Other Adverse Events (participants affected / at risk) | 189/203 | 66/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A: Standard Vincristine Dosing (N=203) | Arm B: Randomized High Dose Vincristine Regimen (N=68)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death NOS (General disorders) | 15 (15) | 1 (1)
Edema face (General disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 2 (2) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 2 (2) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 7 (9) | 6 (7)
Lung infection (Infections and infestations) | 2 (2) | 1 (1)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 8 (8) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (3) | 1 (1)
Platelet count decreased (Investigations) | 3 (3) | 2 (2)
White blood cell decreased (Investigations) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 2 (2)
Myelitis (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 4 (4) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A: Standard Vincristine Dosing (N=203) | Arm B: Randomized High Dose Vincristine Regimen (N=68)
Anemia (Blood and lymphatic system disorders) | 51 (102) | 22 (40)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 127 (250) | 48 (89)
Hemolysis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 4 (4) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Wolff-Parkinson-White syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 1 (2)
Optic nerve disorder (Eye disorders) | 1 (5) | 1 (1)
Photophobia (Eye disorders) | 2 (2) | 1 (1)
Retinopathy (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 14 (16) | 7 (11)
Anal fistula (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anal mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Anal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 9 (10) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 17 (18) | 11 (12)
Duodenal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 43 (53) | 17 (27)
Nausea (Gastrointestinal disorders) | 7 (7) | 6 (7)
Oral pain (Gastrointestinal disorders) | 3 (4) | 6 (9)
Pancreatitis (Gastrointestinal disorders) | 10 (11) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal mucositis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 6 (7) | 1 (1)
Vomiting (Gastrointestinal disorders) | 15 (16) | 6 (6)
Edema limbs (General disorders) | 2 (2) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (2)
Fever (General disorders) | 32 (37) | 4 (4)
Flu like symptoms (General disorders) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (2) | 0 (0)
Infusion related reaction (General disorders) | 2 (2) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0)
Localized edema (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 9 (9) | 7 (7)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 5 (5) | 0 (0)
Anaphylaxis (Immune system disorders) | 10 (12) | 7 (8)
Immune system disorders - Other, specify (Immune system disorders) | 0 (0) | 1 (1)
Anorectal infection (Infections and infestations) | 3 (3) | 1 (1)
Appendicitis (Infections and infestations) | 5 (5) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (2)
Bladder infection (Infections and infestations) | 3 (3) | 0 (0)
Bone infection (Infections and infestations) | 2 (2) | 0 (0)
Bronchial infection (Infections and infestations) | 3 (3) | 0 (0)
Catheter related infection (Infections and infestations) | 30 (35) | 3 (4)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 9 (9) | 5 (7)
Eye infection (Infections and infestations) | 0 (0) | 1 (1)
Hepatic infection (Infections and infestations) | 2 (2) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 101 (207) | 47 (135)
Joint infection (Infections and infestations) | 1 (1) | 0 (0)
Lip infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 22 (27) | 7 (8)
Lymph gland infection (Infections and infestations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 5 (5) | 0 (0)
Otitis media (Infections and infestations) | 4 (5) | 0 (0)
Pancreas infection (Infections and infestations) | 1 (3) | 0 (0)
Paronychia (Infections and infestations) | 3 (4) | 0 (0)
Penile infection (Infections and infestations) | 1 (1) | 0 (0)
Peripheral nerve infection (Infections and infestations) | 2 (2) | 0 (0)
Pleural infection (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 25 (32) | 4 (4)
Sinusitis (Infections and infestations) | 4 (5) | 2 (3)
Skin infection (Infections and infestations) | 16 (16) | 2 (2)
Soft tissue infection (Infections and infestations) | 2 (2) | 1 (1)
Upper respiratory infection (Infections and infestations) | 9 (9) | 1 (1)
Urinary tract infection (Infections and infestations) | 13 (17) | 3 (3)
Wound infection (Infections and infestations) | 5 (6) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 5 (5) | 4 (4)
Alanine aminotransferase increased (Investigations) | 79 (153) | 24 (43)
Alkaline phosphatase increased (Investigations) | 3 (5) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 54 (74) | 18 (24)
Blood bilirubin increased (Investigations) | 15 (18) | 10 (10)
Cholesterol high (Investigations) | 4 (5) | 0 (0)
Creatinine increased (Investigations) | 4 (4) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
Fibrinogen decreased (Investigations) | 8 (8) | 4 (4)
GGT increased (Investigations) | 12 (16) | 2 (4)
INR increased (Investigations) | 0 (0) | 1 (1)
Investigations - Other, specify (Investigations) | 2 (2) | 0 (0)
Lipase increased (Investigations) | 17 (19) | 4 (4)
Lymphocyte count decreased (Investigations) | 15 (34) | 5 (9)
Neutrophil count decreased (Investigations) | 127 (421) | 44 (152)
Platelet count decreased (Investigations) | 93 (201) | 32 (72)
Serum amylase increased (Investigations) | 11 (13) | 3 (4)
Weight gain (Investigations) | 1 (1) | 1 (1)
Weight loss (Investigations) | 3 (3) | 1 (1)
White blood cell decreased (Investigations) | 61 (174) | 25 (70)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 20 (23) | 10 (18)
Dehydration (Metabolism and nutrition disorders) | 14 (16) | 7 (9)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 26 (35) | 12 (13)
Hyperkalemia (Metabolism and nutrition disorders) | 8 (9) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypernatremia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 11 (17) | 2 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 19 (21) | 7 (9)
Hypocalcemia (Metabolism and nutrition disorders) | 20 (23) | 8 (15)
Hypokalemia (Metabolism and nutrition disorders) | 63 (103) | 20 (35)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 31 (40) | 12 (15)
Hypophosphatemia (Metabolism and nutrition disorders) | 20 (22) | 4 (4)
Iron overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (11)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7) | 7 (11)
Ataxia (Nervous system disorders) | 1 (1) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Encephalopathy (Nervous system disorders) | 2 (2) | 2 (3)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 5 (9)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 2 (2) | 2 (2)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 9 (11) | 7 (11)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (15) | 10 (19)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 3 (3) | 0 (0)
Syncope (Nervous system disorders) | 7 (7) | 3 (3)
Tremor (Nervous system disorders) | 1 (1) | 1 (1)
Trigeminal nerve disorder (Nervous system disorders) | 0 (0) | 2 (2)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2)
Confusion (Psychiatric disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 4 (5)
Hallucinations (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Personality change (Psychiatric disorders) | 0 (0) | 1 (3)
Psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 6 (6) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 (2) | 2 (2)
Renal calculi (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 20 (25) | 11 (14)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Social circumstances - Other, specify (Social circumstances) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 2 (2) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 4 (5) | 5 (6)
Hypotension (Vascular disorders) | 31 (36) | 9 (9)
Thromboembolic event (Vascular disorders) | 8 (11) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.